CLINICAL TRIAL: NCT00074932
Title: Expanded Access Use of Myozyme (Alglucosidase Alfa) in Patients With Late-onset Pompe Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU02603
Expanded Access: Available
Record Dates: First submitted 2003-12-23; First posted 2003-12-25 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Glycogen Storage Disease Type II; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease; Acid Maltase Deficiency Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Other)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg
  Other Names: Alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The objective of this protocol is to provide enzyme replacement therapy with alglucosidase alfa on an expanded access basis, to severely affected patients with late-onset Pompe disease for whom there is no alternative treatment and who do not meet the clinical characteristics described in the inclusion criteria for participation in other Genzyme Corporation-sponsored studies currently enrolling patients with late-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient or the patient's legal guardian(s) must provide written informed consent prior to any study-related procedures being performed.
* The patient has/had onset of symptoms compatible with Pompe disease after 12 months of age. Age at onset of symptoms must be documented in the patient's medical record(s).
* The patient has documented GAA deficiency consistent with a diagnosis of Pompe disease, or the patient has a confirmed diagnosis of Pompe disease by documented genotype. Tissues used for determination of GAA deficiency may include blood, muscle or skin fibroblasts.
* The patient must have the following conditions: a. The patient must be wheelchair bound (unable to ambulate with the use of assistive devices, such as walker, cane, or crutches) AND b. The patient requires the use of invasive ventilation (defined as the use of any form of ventilatory support applied through an endotracheal tube).
* Female patients of childbearing potential must have a documented negative pregnancy test prior to dosing each month. In addition, all female patients of childbearing potential must use a medically accepted method of contraception throughout the program. Male patients who are sexually active must use a barrier method of contraception.

Exclusion Criteria:

* Use of any investigational product within 30 days prior to program enrollment.
* Major congenital abnormality;
* Clinically significant organic disease (with the exception of symptoms relating to late-onset Pompe disease), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival.
* The patient meets the clinical characteristics described in the inclusion criteria for participation in other Genzyme Corporation-sponsored treatment study currently enrolling patients with late-onset Pompe disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-11; Primary Completion 2006-08 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Provide ERT with Myozyme in severly affected patients with Late-onset Pompe disease | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - Colorado Health Science Center, Aurora, Colorado
  - Galichia Heart Hospital, Wichita, Kansas
  - Genzyme Medical Information, Cambridge, Massachusetts
  - Freeman Health Systems, Joplin, Missouri
  - The Women's and Children's Hospital of Buffalo, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Macoumb/Oakland Adult Medicine, Rochester Hills, New York
  - Riverside Regional Medical Center, Newport News, Virginia